CLINICAL TRIAL: NCT00405327
Title: A Pilot Study of Tumor Lysate-pulsed Dendritic Cell Vaccine for Immune Augmentation for High-risk Solid Tumor Patients Following Autologous Stem Cell Transplantation
Brief Title: A Pilot Study of Tumor Cell Vaccine for High-risk Solid Tumor Patients Following Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Principal Investigator, James Geiger, MD, Professor of Surgery, Pediatric Surgery Section, University of Michigan Rogel Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2005.050; GCRC ID # 2191; HUM00002650 (Other: University of Michigan Medical School)
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Sarcoma; Neuroblastoma; Wilm's Tumor
Keywords: tumor vaccine; metastatic solid tumors; recurrent tumors
MeSH Terms: conditions — Sarcoma; Neuroblastoma; Wilms Tumor; Neoplasms | interventions — Vaccines; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DC vaccine therapy (Experimental): Tumor lysate-pulsed dendritic cell (DC) vaccine following HSCT
  Interventions: Biological: Tumor lysate-pulsed dendritic cell (DC) vaccine; Other: Hematopoietic stem cell transplantation (HSCT)

INTERVENTIONS:
Biological: Tumor lysate-pulsed dendritic cell (DC) vaccine — Tumor lysate-pulsed dendritic cell vaccine
Other: Hematopoietic stem cell transplantation (HSCT) — Hematopoietic stem cell transplantation (HSCT)

SUMMARY:
Localized solid tumors such as, sarcoma, neuroblastoma, and Wilms' tumor, can generally be effectively treated with a combination of surgery, radiation and chemotherapy. However, patients with metastatic or relapsed disease have a very poor prognosis.

New approaches to the management of these difficult groups of patients are needed. There is evidence to suggest that solid tumors may be good candidates for immunotherapy approaches. In fact, recent experimental evidence indicates that the period of lymphopenia that occurs after stem cell transplant may be an opportune time to use an immunotherapy treatment approach. In light of the very poor prognosis of young patients with advanced solid tumors, this treatment approach warrants further investigation.

DETAILED DESCRIPTION:
Localized solid tumors such as, sarcoma, neuroblastoma, and Wilms' tumor, can generally be effectively treated with a combination of surgery, radiation and chemotherapy. However, patients with metastatic or relapsed disease have a very poor prognosis.

For the past decade, efforts to increase overall survival and progression-free survival for patients with high-risk pediatric and young adult tumors, have evaluated the use of high-dose chemotherapy and hematopoietic stem cell transplantation (HSCT). The proportion of patients who enter a complete remission with HSCT is high, ranging from 81 to 90%. While autologous HSCT renders a large proportion of patients temporarily disease-free, relapse develops in the majority of patients.

Survival appears to have been most improved with this strategy for neuroblastoma, but relapses occur in the majority of patients. Similar strategies have also been tried for patients with advanced stage sarcoma and Wilms' tumor, but relapses are even more problematic.

New approaches to the management of these difficult groups of patients are needed. There is evidence to suggest that solid tumors may be good candidates for immunotherapy approaches. In fact, recent experimental evidence indicates that the period of lymphopenia that occurs after HSCT may be an opportune time to use this treatment approach. In light of the very poor prognosis of young patients with advanced solid tumors, this treatment approach warrants further investigation.

ELIGIBILITY:
Eligibility

Inclusion Criteria:

To participate in this study, it is necessary to collect sufficient tumor and peripheral blood stem cells to both develop the vaccine and perform the autologous stem cell transplant. Patients who also have previously had tumor or stem cells collected, which are available and sufficient for this study, are eligible to participate as study subjects.

1. Patients must have a histologically verified diagnosis of neuroblastoma, Wilm's tumor, or sarcoma, including rhabdomyosarcoma, a Ewing's sarcoma family tumor (ES, PNET), synovial sarcoma, fibrosarcoma, or desmoplastic round cell tumor.

   and must meet one of the following criteria:
   1. have metastatic disease at diagnosis
   2. have never achieved complete remission following frontline standard therapy
   3. have relapsed after receiving standard therapy
2. Patients must have been < 30 years of age at the time of original diagnosis.
3. Patients must have a source of tumor tissue from which approximately 1 gram of viable tumor can be obtained for vaccine development.
4. Patients must have a good performance status (>70% by Lansky or Karnofsky scales).
5. Patients must have a life expectancy of at least 16 weeks.
6. Females of child-bearing age (>= 12 years old) must have a negative pregnancy test.

   Patients may enroll on this study at various points in their treatment including diagnosis, recurrence, or just prior to initiation of study mandated transplant therapy. Because patients may enter this study prior to completion of retransplant treatments, the below criteria must be met only to proceed to the high dose chemotherapy and autologous stem cell transplant part of this study. These criteria are not a requirement to enter this study in order to collect tumor or peripheral blood stem cells.
7. Patients must have achieved complete response or very good partial response(>= 90% decrease in tumor volume) before proceeding to transplant. For patients enrolling on this study just prior to transplant a VGPR or CR must be achieved to be eligible.
8. Patients may have undergone prior autologous peripheral blood stem cell transplantation, provided at least 12 months have elapsed prior to entry on this study.
9. Patients must have had a successful peripheral blood stem cell collection, with cryopreservation of PBSCs for both engraftment and for generation of dendritic cells.
10. Adequate baseline organ function must be present:

    hematologic parameters (not applicable if bone marrow is involved with tumor):
    1. ANC > 500/mm3
    2. platelet count > 50,000/mm3
    3. serum creatinine < 1.5x upper limit of normal for age
    4. serum hepatic transaminases (AST, ALT) < 3x upper limit of normal
    5. serum bilirubin < 1.5x upper limit of normal
    6. cardiac echocardiogram with either SF > 27% or EF > 50%. A comparable EF on a MUGA scan will also meet eligibility criteria.
11. Give or obtain informed consent

Exclusion Criteria:

1. Patients who have received prior antitumor vaccines are ineligible
2. Patients who meet the response criteria but progress prior to study enrollment are ineligible
3. Patients with known autoimmune diseases or conditions are ineligible
4. Patients with HIV infection, AIDS, hepatitis B surface antigen positivity, ongoing bleeding, or any significant uncontrolled medical or psychiatric illness are ineligible.
5. Patients under treatment for infection must cleared by BMT physician prior to enrollment.
6. Patients who are pregnant or nursing are ineligible
7. Prior allogenic transplant

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2006-06; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To estimate the rate of immune response of this immunotherapy treatment | 70 days

SECONDARY OUTCOMES:
To correlate and characterize the immune response to the clinical response. | three years
To define immunologic endpoints that can serve as surrogates of clinical response. | three years

CONTACTS AND LOCATIONS:
Overall Officials: James D Geiger, M.D., Principal Investigator — University of Michigan, Department of Surgery, Pediatric Section
Locations (1):
- University of Michigan, Department of Surgery, Pediatric Section, Ann Arbor, Michigan, United States